CLINICAL TRIAL: NCT00128336
Title: The Heat Study: A 2-year Lifestyle Intervention in Overweight Women to Determine Optimal Approaches for Successful Maintenance of Weight Loss
Brief Title: The Heat Study: 2 Year Lifestyle Intervention in Overweight Women to Encourage Weight Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: Edgar National Centre for Diabetes Research (Other)
Responsible Party: Principal Investigator, Rachael Taylor, PhD student, University of Otago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03/173
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Type 2 Diabetes Mellitus
Keywords: Weight; Diet; exercise; maintenance
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2; Body Weight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nurse support (Active Comparator)
  Interventions: Behavioral: Lifestyle: diet and exercise intervention
- Intensive support (Experimental)
  Interventions: Behavioral: Lifestyle: diet and exercise intervention
- High carbohydrate diet (Active Comparator)
  Interventions: Behavioral: Lifestyle: diet and exercise intervention
- High mono-unsaturated fat diet (Experimental)
  Interventions: Behavioral: Lifestyle: diet and exercise intervention

INTERVENTIONS:
Behavioral: Lifestyle: diet and exercise intervention

SUMMARY:
The purpose of this trial is to determine the most cost effective programme for overweight and obese individuals to maintain weight loss over a 2 year period.

DETAILED DESCRIPTION:
Although short term weight loss is often achievable in overweight individuals, long term maintenance is generally poor. The researchers urgently need new information regarding the most cost effective programme(s) for maintenance of weight loss. This study will recruit 200 women and compare two approaches for providing support: one with intensive health professional support, the other peer group support facilitated by a research nurse with frequent 'weigh- ins'. The researchers will also compare two different diets one a high carbohydrate, high fibre, low glycaemic index diet versus one relatively high in monounsaturated fat and protein and low in glycaemic load.

ELIGIBILITY:
Inclusion Criteria:

* Female participants
* Aged 25 to 70
* Those who have intentionally lost more than or equal to 5% of initial body weight in the previous 6 months will be recruited
* Objective evidence that volunteers were overweight or obese and have lost weight will be obtained from doctors records

Exclusion Criteria:

* Presence of major illness including cancers
* Established cardiovascular disease or stroke
* Diabetes
* Gestational diabetes
* Renal disease
* Malabsorption disorders
* Thyroid disorders
* Major psychiatric disorders
* Taking weight loss medication or medications known to cause weight gain
* Planning a pregnancy in the next 2 years
* Those who do not intend to be in the area for the next 2 years

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Weight | 2 years

SECONDARY OUTCOMES:
Body composition | 2 years
Waist circumference and blood pressure | 2 years
Lipid profile and glucose and insulin | 2 years
Dietary intake | 2 years
Physical fitness | 2 years
Change in mood state | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kelly S Whiteford, MSc (Dist), Principal Investigator — University of Otago
Locations (1):
- Department of Human Nutrition, University of Otago, Dunedin, New Zealand

REFERENCES:
- [Derived] Dale KS, McAuley KA, Taylor RW, Williams SM, Farmer VL, Hansen P, Vorgers SM, Chisholm AW, Mann JI. Determining optimal approaches for weight maintenance: a randomized controlled trial. CMAJ. 2009 May 12;180(10):E39-46. doi: 10.1503/cmaj.080974. PMID 19433812